CLINICAL TRIAL: NCT07044011
Title: Study on Precise Phenotyping Classification in Atrial Fibrillation
Brief Title: Precise Phenotyping Classification in Atrial Fibrillation
Acronym: PPC-AF
Status: Not yet recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Ligang Ding, Professor, China National Center for Cardiovascular Diseases
Other Study IDs: T2022-ZX016
Record Dates: First submitted 2025-06-09; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation, classification
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial fibrillation group: Patients with atrial fibrillation

SUMMARY:
This study aims to integrate multi-omics data (genomics, imaging, serology, etc.) to achieve precise phenotyping classification for atrial fibrillation (AF) patients and explore personalized rhythm control strategies. By enrolling over 1,000 AF patients, we will collect genomic data including GWAS and single-cell sequencing, combined with cardiac MRI, CT, echocardiography imaging, and serum biomarkers, to uncover AF pathological mechanisms and recurrence risks at molecular and structural levels. Machine learning and AI algorithms will be employed to develop AF phenotypic classification models, which will be validated across multiple centers to assess their accuracy and reliability in predicting AF recurrence and therapeutic responses. Furthermore, clinical trials will evaluate the efficacy of oral dronedarone hydrochloride tablets and intravenous nicorandil hydrochloride in preventing post-catheter ablation recurrence and their safety/effectiveness in early cardioversion. Finally, based on advanced phenotyping results, we will establish personalized rhythm control strategies integrating pharmacotherapy, catheter ablation, and lifestyle interventions to optimize AF management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with atrial fibrillation.
2. Voluntarily participated in the study and signed the informed consent form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with atrial fibrillation.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia | 1 year after catheter ablation of atrial fibrillation.
  Atrial arrhythmia events lasting more than 30 seconds within 3 months to 1 year after catheter ablation of atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Van Gelder IC, Rienstra M, Bunting KV, Casado-Arroyo R, Caso V, Crijns HJGM, De Potter TJR, Dwight J, Guasti L, Hanke T, Jaarsma T, Lettino M, Lochen ML, Lumbers RT, Maesen B, Molgaard I, Rosano GMC, Sanders P, Schnabel RB, Suwalski P, Svennberg E, Tamargo J, Tica O, Traykov V, Tzeis S, Kotecha D; ESC Scientific Document Group. 2024 ESC Guidelines for the management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2024 Sep 29;45(36):3314-3414. doi: 10.1093/eurheartj/ehae176. No abstract available. PMID 39210723
- [Background] Tzeis S, Gerstenfeld EP, Kalman J, Saad EB, Shamloo AS, Andrade JG, Barbhaiya CR, Baykaner T, Boveda S, Calkins H, Chan NY, Chen M, Chen SA, Dagres N, Damiano RJ, De Potter T, Deisenhofer I, Derval N, Di Biase L, Duytschaever M, Dyrda K, Hindricks G, Hocini M, Kim YH, la Meir M, Merino JL, Michaud GF, Natale A, Nault I, Nava S, Nitta T, O'Neill M, Pak HN, Piccini JP, Purerfellner H, Reichlin T, Saenz LC, Sanders P, Schilling R, Schmidt B, Supple GE, Thomas KL, Tondo C, Verma A, Wan EY. 2024 European Heart Rhythm Association/Heart Rhythm Society/Asia Pacific Heart Rhythm Society/Latin American Heart Rhythm Society expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2024 Sep;21(9):e31-e149. doi: 10.1016/j.hrthm.2024.03.017. Epub 2024 Apr 8. PMID 38597857